CLINICAL TRIAL: NCT00380094
Title: TRIAGE NOW: Triage in Acute General Chest Pain Patients Evaluation
Brief Title: Triage Now: an Observational, Prospective Multimarker Study of Biomarkers in Patients Presenting With Chest Pain
Status: Completed | Type: Observational
Sponsor: Abbott RDx Cardiometabolic (Other)
Other Study IDs: 0024
Record Dates: First submitted 2006-09-21; First posted 2006-09-25 (Estimated); Last update posted 2009-12-18 (Estimated); Status verified 2009-12

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction
Keywords: ACS; NSTEMI; Myeloperoxidase; nonST segment elevation myocardial infarction
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Study of diagnostic tests for heart attack for patients with chest pain.

DETAILED DESCRIPTION:
Study of multiple biomarkers, including myeloperoxidase, in the evaluation of patients presenting with suspected acute coronary syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Chest pain and ACS in differential diagnosis
* Age> 18 years
* Ability to give informed consent

Exclusion Criteria:

* Trauma
* Vulnerable populations
* Known inflammatory condition

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with chest pain and ACE in differential diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2006-08; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Blankenberg, MD, Principal Investigator — Johannes Gutenberg University Mainz
Locations (1):
- University of Mainz, Mainz, Germany